CLINICAL TRIAL: NCT04298138
Title: Phase One, Open Label Assessment of a Dengue-3-Virus-Live Virus Human Challenge - (DENV-3-LVHC) Virus Strain
Brief Title: Dengue 3 Human Infection Model (DENV-3)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 2019-01-UMU
Record Dates: First submitted 2020-02-21; First posted 2020-03-06 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2022-06

CONDITIONS: Dengue
Keywords: Dengue; Flavivirus Infections; Virus Diseases
MeSH Terms: conditions — Dengue; Flavivirus Infections; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Nine subjects will be assigned to the low dose group. Twenty-one days post inoculation, data will be reviewed for safety and if performance parameters are met. If safety profile is acceptable but performance parameters have not been met, dose escalation to the medium dose will proceed in nine additional subjects. Twenty-one days post middle dose inoculation, data will be reviewed as above and a determination will be made to proceed to the high dose.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose DENV-3-LVHC (Experimental): Dengue-3 Virus-Live Virus Human Challenge (DENV-3-LVHC) single low dose (0.5 mL of 1.4 x 10^3 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously
  Interventions: Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC)
- Medium dose DENV-3-LVHC (Experimental): Dengue-3 Virus-Live Virus Human Challenge (DENV-3-LVHC) single medium dose (0.5 mL of 1.4 x 10^4 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously
  Interventions: Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC)
- High dose DENV-3-LVHC (Experimental): Dengue-3 Virus-Live Virus Human Challenge (DENV-3-LVHC) single high dose (0.5 mL of 1.4 x 10^5 plaque forming units/milliliter (PFU/mL) inoculated subcutaneously
  Interventions: Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC)

INTERVENTIONS:
Biological: Dengue virus 3 Live Virus Human Challenge (DENV-3-LVHC) — Dengue subtype 3 Challenge Virus (DENV-3) strain CH53489 administered as a single injection.

SUMMARY:
To evaluate the effectiveness of candidate dengue vaccine formulations, it is prudent to develop an appropriate challenge model. This study will examine the safety and effectiveness of the Dengue 3 Live Virus Human Challenge (DENV-3-LVHC) product and assess the ability of this virus strain to elicit an uncomplicated dengue-like illness.

DETAILED DESCRIPTION:
Healthy subjects between 18 and 45 years old will be inoculated with Dengue 3 Live Virus Human Challenge (DENV-3-LVHC) in a dose ranging study. Subjects will be closely monitored for the first 28 days with continued follow up through 6 months. Clinical and laboratory parameters, viremia and antibody levels will be assessed. The goal is to determine the dose that produces uncomplicated dengue-like illness.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-45 at the time of consent
2. Ability and willingness to sign informed consent
3. Passing score on comprehension test of at least 75%, with up to 3 attempts
4. Available for the study period
5. Willing to use contraception for the duration of the study
6. Provide consent for release of medical history records from primary care physician, college or university, urgent care or emergency room visit

Exclusion Criteria:

1. Female: pregnant or lactating
2. Heavy menstrual bleeding within the last 6 months- menstrual periods lasting longer than 6 days, or requiring 5 or more pads or tampons per day.
3. Female subjects using an intrauterine device (IUD) or Mirena®
4. Female subjects with fibroids or uterine polyps, endometriosis, adenomyosis, and uterine scarring (e.g., after D&C)
5. Blood tests confirming infection with human immunodeficiency virus- 1 (HIV-1), hepatitis C, hepatitis B (assessed by HbsAg) virus, or positive antibodies to the flaviviruses (FV) dengue, West Nile, Yellow Fever, Japanese encephalitis, or Zika.
6. Active Diabetes or active peptic ulcer disease (PUD)
7. Chronic obstructive pulmonary disease (COPD) or coronary artery disease (CAD)
8. Known or suspected congenital or acquired immunodeficiency; or receipt of immunomodulation therapy such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months)
9. Current, or a history of, auto-immune disease
10. History of Guillain-Barré syndrome (GBS)
11. Any history of FV infection or FV vaccination; or planned FV vaccination, outside the study protocol, during the study period
12. Diagnosis with Bipolar Disorder or Schizophrenia, hospitalization in the past year for a mental health disorder, or any other psychiatric condition, which in the opinion of the investigator prevents the subject from participating in the study.
13. Planned travel during the study period (180 days) which would interfere with the ability to complete all study visits
14. Recent (in the past 4 weeks) travel to any dengue endemic area. These potential subjects may be eligible for enrollment a minimum of 4 weeks later
15. Any laboratory abnormalities prior to inoculation for the tests specified in Table 18 and Table 19 of the protocol, that are considered by the investigator to be clinically significant except those listed in exclusion criteria 16
16. Subjects with the following grade 2 or greater lab abnormalities: Creatinine; Liver Function Tests - ALT, AST; Hemoglobin (females and males); White Blood Cell (WBC) decrease; Platelets decreased; Prothrombin Time (PT); Partial Thromboplastin Time (PTT); Fibrinogen decrease
17. Significant screening physical examination abnormalities at the discretion of the investigator
18. Women who intend to become pregnant or men who intend to father a child during the study period (approximately 180 days)
19. Hives, shortness of breath, swelling of the lips or throat, or hospitalization related to a previous vaccination or an allergy to specific medications/animals for which antigens may be in the virus preparations to include: shellfish allergy, fetal bovine serum, L-glutamine, neomycin and streptomycin
20. Planning to donate blood in the 1 year following inoculation with dengue
21. Recent blood donation within prior 56 days of inoculation
22. Receipt of blood products or antibodies within 56 days of inoculation or during the study period
23. Participation (active or follow-up phase) or planned participation in another vaccine, drug, medical device, or medical procedure clinical trial in the 4 weeks prior to this trial, during the trial, or 6 months following inoculation in this clinical trial
24. Recent or scheduled receipt of any vaccine 4 weeks prior to or after virus inoculation
25. Beliefs that bar the administration of blood products or transfusions
26. Positive urine screen for cocaine, amphetamines, or opiates
27. Currently taking Methadone or Suboxone
28. Currently taking anti-coagulant medication, aspirin or non-steroidal anti-inflammatory drugs (NSAIDs)
29. Chronic migraine headaches, defined as more than 15 headache days per month over a 3-month period of which more than 8 are migraines, in the absence of medication over use
30. Chronic medical condition that, in the opinion of the investigator, impacts subject safety.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Number of Abnormal Laboratory Measurements | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Total number of all abnormal labs
Intensity of Abnormal Laboratory Measurements | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Graded according clinical laboratory normals and FDA toxicity scale
Duration of Abnormal Laboratory Measurements | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of days of abnormal lab
Occurrence of Solicited Injection Site Symptoms | 7 days post virus inoculation
  Number of solicited symptoms
Intensity of Solicited Injection Site Symptoms | 7 days post virus inoculation
  Graded according to FDA toxicity scale
Duration of Solicited Injection Site Symptoms | 7 days post virus inoculation
  Number of days per symptom
Occurrence of Unsolicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of unsolicited site symptoms
Intensity of Unsolicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Graded according to FDA toxicity scale
Duration of Unsolicited Injection Site Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of days per symptom
Occurrence of Solicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of solicited systemic symptoms
Intensity of Solicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Graded according to FDA toxicity scale
Duration of Solicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of days per symptom
Occurence of Unsolicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of unsolicited systemic symptoms
Intensity of Unsolicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Graded according to FDA toxicity scale
Duration of Unsolicited Systemic Symptoms | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Number of days per symptom
Number of Serious Adverse Events | 28 days post virus inoculation or 7 days post hospitalization, whichever is later
  Total number
Number of Serious Adverse Events | 6 months post virus inoculation
  Total number

SECONDARY OUTCOMES:
Incubation period before onset of fever | Up to 28 days post virus inoculation
  Number of days prior to fever
Viremia by Reverse Transcriptase-Polymerase Chain Reaction (RT-PCR) | Up to 28 days post virus inoculation
  Levels of viremia
Occurence of fever | Up to 28 days post virus inoculation
  Defined as greater than or equal to 38°C (100.4°F) measured at least 2 times in 24 hours but not lasting more than 72 hours
Occurrence of Headache | Up to 28 days post virus inoculation
  Number of headaches
Grade of Headache | Up to 28 days post virus inoculation
  Graded according to FDA toxicity scale
Occurrence of Myalgia | Up to 28 days post virus inoculation
  Number of reported myalgias
Grade of Myalgia | Up to 28 days post virus inoculation
  Graded according to FDA toxicity scale
Occurrence of Rash | Up to 28 days post virus inoculation
  Number of rashes
Grade of Rash | Up to 28 days post virus inoculation
  Graded according to FDA toxicity scale
Occurrence of Abnormal Liver Function Test [alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] | Up to 28 days post virus inoculation
  Number of abnormal liver function tests
Grade of Abnormal Liver Function Test [alanine aminotransferase (ALT) and aspartate aminotransferase (AST)] | Up to 28 days post virus inoculation
  Graded according clinical laboratory normals and FDA toxicity scale
Occurrence of Leukopenia | Up to 28 days post virus inoculation
  Number of occurrences
Grade of Leukopenia | Up to 28 days post virus inoculation
  Graded according clinical laboratory normals and FDA toxicity scale
Occurrence of Thrombocytopenia | Up to 28 days post virus inoculation
  Number of occurrences
Grade of Thrombocytopenia | Up to 28 days post virus inoculation
  Graded according clinical laboratory normals and FDA toxicity scale

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Thomas, MD, Principal Investigator — State University of New York, Upstate Medical University (SUNY-UMU)
Locations (1):
- State University of New York, Upstate Medical University (SUNY-UMU), Syracuse, New York, United States

IPD SHARING:
Plan to Share IPD: No